CLINICAL TRIAL: NCT05602051
Title: Efficacy of Mindfulness-based Virtual Reality Intervention on the Symptoms Associated With Hematologic Neoplasms Patients During Chemotherapy
Brief Title: Mindfulness-based Virtual Reality Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wu Yuan, master, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-SR-586
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Hematologic Neoplasms
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality+Mindfulness (Experimental): Intervention method combining virtual reality technology and mindfulness therapy, twice a week, lasting for 7 weeks
  Interventions: Device: virtual reality device
- Mindfulness (No Intervention): Intervention method of mindfulness therapy, twice a week, lasting for 7 weeks

INTERVENTIONS:
Device: virtual reality device — mindfulness combined with virtual reality
  Other Names: Mindfulness
  Arms: Virtual reality+Mindfulness

SUMMARY:
Through virtual reality technology and mindfulness therapy, we can intervene the patients with Hematologic Neoplasms during chemotherapy, hoping to improve their symptoms and self-efficacy.

DETAILED DESCRIPTION:
In recent years, the intervention method of giving mindfulness has achieved good results in the management of symptoms related to cancer patients, but the compliance of patients with conventional mindfulness intervention is low. The virtual reality intervention based on mindfulness can effectively mobilize the enthusiasm of patients to participate in research and the compliance of mindfulness training. We aim to combine virtual reality with mindfulness intervention to intervene patients with hematologic neoplasms during chemotherapy, To improve their symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hematologic Neoplasms(leukemia, lymphoma or multiple myeloma) and receiving chemotherapy
* Hospitalized for more than 4 weeks
* Have normal communication ability, clear consciousness, and willing to participate in this study

Exclusion Criteria:

* People are cognitive dysfunction and audio-visual dysfunction
* Have mental problems or have reported mental disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
MDASI-C | up to 7 weeks
  Symptom burden was assessed using the Chinese version of the M. D. Anderson Symptom Inventory (MDASI-C),39 which is a self-report scale consisting of two domains. The first domain is named "core symptom severity items" and has 13 symptoms. Each symptom is rated on an 11-point scale (0-10) to indicate the presence and severity of the symptom, with 0 indicating "not present" and 10 indicating "as bad as you can imagine." Each symptom is rated based on the severity of the symptom, at its worst, in the last 24 h. The second domain is named "six symptoms interference items" and includes ratings of how much symptoms interfered with different aspects of the survivor's life in the last 24 h. The interference items are also rated on a scale of 0-10, with 0 indicating "did not interfere" and 10 indicating "interfered completely." A score of 0-3 indicated a mild level, 4-6 indicated a moderate level, and 7-10 indicated a severe level of symptom severity or interference.
Hospital Anxiety and Depression Scale (HADS) | up to 7 weeks
  The hospital anxiety and depression scale The HADS was compiled by Zigmond AS Which was used to detect states of depression and anxiety in the setting of an hospital medical outpatient clinic . It is a 14-question instrument, with each question being scored between 0 (no impairment) and 3 (severe impairment), with a maximum score of 21 for anxiety or depression.

SECONDARY OUTCOMES:
the self-management efficacy scale (C-SUPPH) | up to 7 weeks
  the self-management efficacy scale (C-SUPPH)，The C-SUPPH scale consisted of 28 items in three dimensions: self-decompression, self-decision-making, and positive attitude, with each item scoring 1-5 points and a total score of 28-140 points. The higher the total score is, the higher the self-efficacy is.

CONTACTS AND LOCATIONS:
Overall Officials: yuxi Zhang, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No